CLINICAL TRIAL: NCT05883371
Title: Investigating Mechanisms of Participatory Autoimmune Condition Treatment (IMPACT): An Outcomes Research Registry of a Comprehensive Approach to Autoimmune Disorders
Brief Title: IMPACT - AndHealth Autoimmune Research Registry
Status: Recruiting | Type: Observational
Sponsor: AndHealth (Industry)
Responsible Party: Sponsor
Other Study IDs: 044-AND
Record Dates: First submitted 2023-05-05; First posted 2023-05-31 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-05

CONDITIONS: Arthritis, Rheumatoid; Arthritis, Psoriatic; Psoriasis; Ankylosing Spondylitis; Autoimmune Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Psoriasis; Spondylitis, Ankylosing; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Root-cause autoimmune treatment program — The AndHealth autoimmune treatment program combines validated and guideline-driven approaches along with emerging evidence-based modalities. The program includes a comprehensive assessment of disease severity, analysis of root causes and comorbidities, and an evaluation of the patient's readiness for implementing important lifestyle changes. This is followed by the development of an optimized and personalized plan to achieve and sustain clinical remission while monitoring their progress. Each patient participating in the AndHealth program receives a personalized care plan developed by the patient's medical provider in collaboration with a team of healthcare specialists. Helping a patient manage everyday lifestyle decisions can have a profound effect on their ability to achieve and maintain remission. The AndHealth Program has organized these into four basic groups of lifestyle behaviors: 1.) Dietary/Nutrition, 2.) Sleep/Circadian, 3.) Stress/HPA axis, and 4.) Physical Activity.

SUMMARY:
This is a patient research registry aimed at evaluating the effectiveness of a comprehensive, root-cause medical approach ("AndHealth program") for autoimmune disorders. This approach involves a combination of pharmacological and non-pharmacological therapies offered under the care of a licensed physician with the support of health coaches. While protocol guidance is provided, the therapeutic approach is personalized to the individual needs of patients. The autoimmune disorders of focus in this registry include rheumatoid arthritis, psoriatic arthritis, psoriasis and ankylosing spondylitis. A variety of validated labs, patient-reported outcomes, and medication usage will be assessed among participating patients over a period of up to five years to evaluate the long-term effectiveness of this approach.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 70 years of age
2. Able to understand and write English
3. Voluntarily consent to the study and understand its nature and purpose including potential risks and side effects
4. Documented diagnosis and current use/recommendation for biologic or DMARD medications to treat rheumatoid arthritis, psoriatic arthritis, psoriasis, or ankylosing spondylitis.

Exclusion Criteria:

1. Pregnant, breastfeeding, or planning to become pregnant in the next 12 months
2. Advanced liver or kidney disease
3. Previous organ transplant or awaiting organ transplant
4. Actively being treated for cancer
5. Poorly-controlled mental illness (i.e., schizophrenia, bipolar, current eating disorder)
6. Has a terminal illness
7. Current opioid use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of AndHealth patients with a documented diagnosis and current use or recommendation for biologic or DMARD medications to treat the autoimmune disorders under study (rheumatoid arthritis, psoriatic arthritis, psoriasis, or ankylosing spondylitis) and who elect to participate in the outcomes research registry.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2023-11-22 (Estimated); Study Completion 2028-05-22 (Estimated)

PRIMARY OUTCOMES:
PROMIS - Global Health | Baseline and approximately quarterly thereafter for up to 5 years
  Change in PROMIS - Global Health is a co-primary outcome for all patients. All patients will provide the PROMIS - Global Health at baseline and all follow-up visits. The 10-item PROMIS Global Health is a patient-reported survey that was designed for use in complex heterogeneous patient populations. The PROMIS Global Health measures overall health status across several physical and mental health areas. PROMIS t-scores range from 16.2 to 67.7 (Physical Health) and 21.2 to 67.6 (Mental Health) with higher scores indicating better health.
Routine Assessment of Patient Index Data 3 (RAPID 3) | Baseline and approximately quarterly thereafter for up to 5 years
  Change in RAPID 3 is a co-primary outcome for rheumatoid arthritis & psoriatic arthritis patients. All patients with rheumatoid and psoriatic arthritis will provide the RAPID 3 at baseline and all follow-up visits. This 3-item questionnaire is a rheumatological disease activity index that is calculated to reflect severity of disease. Scores range from 0 to 30 with higher scores indicating worse symptoms.
Dermatology Life Quality Index (DLQI) | Baseline and approximately quarterly thereafter for up to 5 years
  Change in DLQI is a co-primary outcome for psoriasis patients. All patients with psoriasis and psoriatic arthritis will provide the DLQI at baseline and all follow-up visits. This 10-item questionnaire is a common measure of the health-related quality of life for skin disorders. DLQI scores range from 0 to 30, with higher scores indicating worse quality of life.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline and approximately quarterly thereafter for up to 5 years
  Change in BASDAI is a co-primary outcome for ankylosing spondylitis patients. All patients with ankylosing spondylitis will provide the BASDAI at baseline and all follow-up visits. This 6-item questionnaires is a brief, validated measure of ankylosing spondylitis activity. BASDAI scores range from 0 to 10, with higher scores indicating worse symptoms.

SECONDARY OUTCOMES:
Patient Health Questionnaire for Anxiety and Depression (PHQ4) | Baseline and approximately quarterly thereafter for up to 5 years
  Change in PHQ4 is a secondary outcome for all patients. All patients will provide the PHQ4 at baseline and at follow-up visits, as is warranted by scores. This 4-item questionnaire is a common measure of anxiety and depression symptoms. PHQ4 scores range from 0 to 12, with higher scores indicating worse symptoms.
Disease Activity Score 28 (DAS28) | Baseline and approximately quarterly thereafter for up to 5 years
  Change in DAS28 is a secondary outcome for rheumatoid arthritis patients. The DAS28 is a measure of disease activity in rheumatoid arthritis that will be assessed at baseline and all follow-up visits for participants with rheumatoid arthritis. DAS stands for 'disease activity score' and 28 joints are examined in this assessment. DAS28 scores range from 0 to 9.4, with higher scores indicating worse symptoms.
Psoriasis Area and Severity Index (PASI) | Baseline and approximately quarterly thereafter for up to 5 years
  Change in PASI is a secondary outcome for psoriasis and psoriatic arthritis patients. The PASI is a measure of psoriasis and psoriatic arthritis severity that will be assessed at baseline and all follow-up visits for participants with psoriasis or psoriatic arthritis. This common clinical measure selects a representative area of psoriasis for each body region. The intensity of redness, thickness, and scaling of the psoriasis is assessed by the clinician. PASI scores range from 0 to 72, with higher scores indicating worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Myles Spar, MD, Principal Investigator — AndHealth
Locations (1):
- AndHealth, Columbus, Ohio, United States